CLINICAL TRIAL: NCT04361331
Title: A Randomized, Open, Two-cohort Phase 2 Study of Toripalimab(PD1) Combined With Lenvatnib, or Gemox Chemotherapy Combined With Lenvatinib as First-line Therapy in Patients With Advanced or Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Two-cohort Study of Toripalimab(PD1)+Lenvatnib, or Gemox+Lenvatinib in Advanced Intrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zs-ICC-2020
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cholangiocarcinoma, Intrahepatic
Keywords: intrahepatic Cholangiocarcinoma; Lenvatinib; Gemox chemotherapy; Programmed cell death protein 1 antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: Arm1: toripalimab combined with lenvatinib， Arm 2: lenvatinib combined with Gemox
Masking Description: Random number table grouping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toripalimab combined with lenvatinib (Other): 1. Toripalimab: 240 mg, intravenous infusion, Q3W;
  2. Lenvatinib: 8mg (body weight <60kg) or 12mg (body weight ≥60kg), qd;
  Interventions: Drug: Toripalimab combined with lenvatinib
- Lenvatinib combined with gemox (Other): 1. Lenvatinib: 8mg (body weight <60kg) or 12mg (body weight ≥60kg), qd
  2. Gemox chemotherapy D1: Oxaliplatin 85mg / m2, Gemcitabine 1g / m2 D8: Gemcitabine 1g / m2 Three weeks are a course, a total of 6-8 courses
  Interventions: Drug: Lenvatinib combined with gemox

INTERVENTIONS:
Drug: Lenvatinib combined with gemox — Arm2: Lenvatinib + gemox
  Other Names: gemox chemotherapy
  Arms: Lenvatinib combined with gemox
Drug: Toripalimab combined with lenvatinib — Toripalimab combined with lenvatinib
  Arms: Toripalimab combined with lenvatinib

SUMMARY:
We aim to explore the effects and safety of the two cohorts of toripalimab combined with lenvatinib or gemox combined with lenvatinib as first-line therapy in advanced or unresectable intrahepatic cholangiocarcinoma

DETAILED DESCRIPTION:
For advanced intrahepatic cholangiocarcinoma (ICC) that cannot be surgically removed or accompanied by metastasis, the NCCN guidelines (NCCN guidelines hepatobiliary cancer, 2019) recommend that the current treatment options are limited, mainly recommending gemcitabine combined with platinum-based antitumor drugs (cisplatin, oxaliplatin, etc.) chemotherapy as first-line treatment. Adding targeted drugs can enhance the anti-tumor effect. For those with microsatellite instability, it is recommended to add anti-PD1(programmed cell death protein 1) antibody. Gemox chemotherapy (oxaliplatin + gemcitabine) has been used in the treatment of advanced intrahepatic cholangiocarcinoma, but the efficacy is still not satisfactory. Lenvatinib is a small-molecule multi-kinase inhibitor that is currently approved for first-line treatment of advanced hepatocellular carcinoma. In recent years, the anti-PD1 antibody has shown efficacy in the treatment of primary liver cancer. Lenvatinib combined with anti-PD1 antibody or chemotherapy may have a better effect than single use for advanced ICC. At present, lenvatinib combined with anti-PD1 antibody or lenvatinib combined with Gemox in the first-line treatment of advanced ICC has not been reported.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient must be required to sign an informed consent; 2. Age 18-75 years old, male or female; 3. ECOG performance status score (PS score) 0 or 1 point; 4. Child-Pugh score A; 5. Intrahepatic cholangiocarcinoma confirmed by histopathology; agree to provide previously stored tumor tissue samples or fresh biopsy tumor lesions; 6. Unresectable ICC patients or postoperative ICC recurrence and metastasis, without systematic treatment within 6 months; 7. The functional indicators of vital organs meet the following requirements

  1. Neutrophils ≥1.5 * 109 / L; platelets ≥100 * 109 / L; hemoglobin ≥9g / dl; serum albumin ≥3g/dl;
  2. Thyroid stimulating hormone (TSH) ≤ 1 times the upper limit of normal value(ULN), T3 and T4 are in the normal range;
  3. Bilirubin ≤ 1.5 times ULN; ALT and AST ≤ 3 times ULN;
  4. Serum creatinine ≤ 1.5 times ULN, creatinine clearance rate ≥ 60ml/min (calculated using Cockcroft-Gault formula); 8. Subject has at least 1 measurable lesion (according to RECIST1.1); 9. Non-lactating or pregnant women, contraception during or 3 months after treatment.

Exclusion Criteria:

* 1. Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma and other non-cholangiocarcinoma malignancies; 2. Existing or concurrently suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid cancer; 3. Have used lenvatinib or gemcitabine-based chemotherapy within 6 months or have used PD1 monoclonal antibody and PD-L1 monoclonal antibody treatment; 4. Severe cardiopulmonary and renal dysfunction; 5. Hypertension that is difficult to control by the drug (systolic blood pressure (BP) ≥140 mmHg and / or diastolic blood pressure ≥90 mmHg) (based on the average of ≥3 BP readings obtained from ≥2 measurements); 6. Abnormal blood coagulation function (PT> 14s), have bleeding tendency or are receiving thrombolysis or anticoagulation treatment; 7. HBV DNA> 2000 copies/ml and HCV RNA>1000 after antiviral treatment; 8. Have a history of esophagogastric varices, with significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment; 9. Active infection requiring systemic treatment and treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, have not received regular anti-TB treatment or tuberculosis Still in the active period; 10. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive; 11. Have a history of psychotropic substance abuse, alcohol or drug abuse; 12. Known to have a history of severe allergies to any monoclonal antibodies, anti-angiogenic targeted drugs, and platinum or gemcitabine; 13. Other factors that may affect the safety of subjects or test compliance as judged by the investigator. Such as serious illness (including mental illness) requiring combined treatment, severe laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  Objective response rate of advanced and unresectable intrahepatic cholangiocarcinoma

SECONDARY OUTCOMES:
Safety: the potential side effects | 12 months
  The potential side effects
Overall survival | 12 months
  From the beginning date of combined therapy to the date of death
Progression free survival | 12 months
  From the beginning date of combined therapy to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD & PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - Zhongshan hospital, Shanghai, Shanghai Municipality
  - Huang xiaoyong, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre T, Tournigand C, Rosmorduc O, Provent S, Maindrault-Goebel F, Avenin D, Selle F, Paye F, Hannoun L, Houry S, Gayet B, Lotz JP, de Gramont A, Louvet C; GERCOR Group. Gemcitabine combined with oxaliplatin (GEMOX) in advanced biliary tract adenocarcinoma: a GERCOR study. Ann Oncol. 2004 Sep;15(9):1339-43. doi: 10.1093/annonc/mdh351. PMID 15319238
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Derived] Huang XY, Shi GM, Zheng ZT, Sun HC, Liang F, Ji Y, Chen Y, Yang GH, Hu ZQ, Lu JC, Meng XL, Guo XJ, Zhang CC, Fan J, Zhou J. Anti-PD1 antibody toripalimab combined with lenvatinib, or GEMOX chemotherapy combined with lenvatinib as first-line therapy in patients with advanced intrahepatic cholangiocarcinoma: a randomized, open, two-cohort Phase 2 Study. BMC Med. 2025 Oct 21;23(1):573. doi: 10.1186/s12916-025-04404-4. PMID 41121202